CLINICAL TRIAL: NCT06250530
Title: Do Patient Specific Implants Improve Accuracy of Correction With MOWHTO. A Pilot Study for a Definitive Randomised Trial Comparing TOMOFIX and BodyCAD Fine Osteotomy.
Brief Title: Comparison Between TOMOFIX and BodyCAD Fine Osteotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Al Getgood, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB #120983
Record Dates: First submitted 2023-12-20; First posted 2024-02-09 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Osteotomy; Malalignment, Bone; Osteoarthritis, Knee
MeSH Terms: conditions — Bone Malalignment; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The proposed study is a single centre, pilot randomised controlled, patient blinded study that will randomly assign 40 participants with medial knee osteoarthritis undergoing medial opening wedge proximal tibial osteotomy (MOWHTO) to either current standard of care, with TOMOFIX plating system, or utilise patient specific instrumentation and custom-made plate development, with BodyCAD Fine Osteotomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BodyCAD (Experimental): For participants randomized to BodyCAD Fine osteotomy, the HKA radiographs and CT scans will be sent to the manufacturer via a secure weblink as per SoC. The films will be used to calculate the desired correction and the instruments and implants manufactured accordingly. The mechanical medial proximal tibial angle (mMPTA) will be recorded for both pre- and planned post-operative situations and used to determine the accuracy of correction (primary outcome).
  Interventions: Procedure: High tibial osteotomy using BodyCAD
- TOMOFIX (Active Comparator): For participants randomized to the TOMOFIX system, preoperative planning will use the HKA radiograph. DICOM images will be transported to MEDICAD software program in which alignment angles and alignment correction will be calculated. The mMPTA will again be utilised to determine the accuracy of correction (primary outcome). The preop CT scan will also be used as per the BodyCAD system and the same indices calculated so as to minimise measurement bias between two different imaging modalities. However, the results of the preoperative 3D CT planning will not be made available to the operating surgeon, again to minimise bias between groups.
  Interventions: Procedure: High tibial osteotomy using TOMOFIX

INTERVENTIONS:
Procedure: High tibial osteotomy using TOMOFIX — TOMOFIX: A guidepin is placed to determine the level and length of the osteotomy with an appropriate hinge position selected. The oscillating saw is then used along with osteotomes to complete the osteotomy under image intensifier guidance. This is opened to the desired width of correction with a trapezoidal gap noted when using laminar spreader in the posterior position to avoid slope change. The plate is then applied and secured as per manufacturers operative technique.
  Other Names: TOMOFIX
  Arms: TOMOFIX
Procedure: High tibial osteotomy using BodyCAD — BodyCAD: The patient specific cutting block is applied to the proximal tibia and secured in placed. The osteotomy is then created with sequential drills and osteotome and opened to the predetermined correction as per the manufacturer's guidelines. The plate is applied and secured with the supplied screws.
  Other Names: BodyCAD
  Arms: BodyCAD

SUMMARY:
This is a single centre, randomised, patient blinded pilot study that will assign 40 participants with medial knee osteoarthritis undergoing medial opening wedge high tibial osteotomy (MOWHTO) to either current standard of care with TOMOFIX plating system, or utilise patient specific instrumentation and custom-made plate development, with BodyCAD Fine Osteotomy. If the definitive study is deemed feasible, an additional 110 participants will be randomized, for a total of 150 participants.

DETAILED DESCRIPTION:
The proposed study is a single centre, pilot randomised controlled, patient blinded study that will randomly assign 40 participants with medial knee osteoarthritis undergoing medial opening wedge proximal tibial osteotomy (MOWHTO) to either current standard of care, with TOMOFIX plating system, or utilise patient specific instrumentation and custom-made plate development, with BodyCAD Fine Osteotomy. Participants will follow a standardized rehabilitation protocol. Outcomes will be assessed over two years postoperatively utilising CT assessment for accuracy of correction, bony union and construct stability as well as PROMs including KOOS and EQ5D.

Complications, adverse events, returns to theatre and costs will also be recorded. End of study is defined when the last enrolled subject reaches the 24-month follow-up time point and close-out activities are complete.

If the pilot study demonstrates the feasibility of the definitive trial, an additional 110 participants will be ennrolled, for a total of 150 participants.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years old
* have medial compartment osteoarthritis, with varus alignment, deemed suitable for a MOWHTO
* able to speak, read and understand English

Exclusion Criteria:

* found to have a cruciate ligament deficiency
* require multiplanar or rotational alignment correction
* have greater than 5 degrees fixed flexion deformity
* unable to have CT scans for follow up
* evidence of tricompartmental osteoarthritis
* evidence of lateral compartment osteoarthritis on arthroscopy
* received injection therapy within 3 months of surgery on the operative knee
* have a medical history of inflammatory arthropathy, diabetes
* actively smoke

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
KOOS | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months
  The KOOS is a 42-item knee-specific questionnaire with five separately reported domains, including pain, other symptoms, function in daily living, function in sports/recreation and knee-related quality of life. Domain scores represent the average of all items in the domain standardized to a score from 0 to 100 (worst to best). This instrument has demonstrated construct validity, excellent test-retest reliability for each domain (range, 0.75 to 0.93) and is responsive to change.

SECONDARY OUTCOMES:
EQ-5D (Index and VAS) | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months
  The EuroQoL comprises two sections, the EQ-5D index and the EQ-5D visual analogue scale (VAS). The EQ-5D index is a 5-item standardized generic measure of HRQOL that includes domains of mobility, self-care, usual activities, pain and discomfort and anxiety and depression. Each item is scored using a 5-point response scale and each combination of response choices describes a health state (3125 unique health states). Each health state can be converted to a utility value from 0 (worst) to 1.0 (best) using a scoring formula. The EQ-5D VAS is a 0 (worst) to 100 (best) scale that assesses patient-perceived health status responsiveness among patients undergoing knee arthroscopy.
Procedure Time | Surgery
  To determine the length of the surgery, the timing will be extracted from the intra-operative nursing record, the time of first incision and the time of closing and calculate the amount of time in minutes. To determine the amount of fluoroscopic time, the time will be extracted from image intensifier record the amount of fluoroscopic imaging utilised in the operating room and calculate a total exposure time in seconds.
Adverse Events | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months
  All adverse events will be recorded and the relatedness, severity and expectedness to the study protocol will be classified. Plain radiographs will be used at each follow-up to assess for the presence of a hinge fracture and delayed or non-union. Loss of motion/arthrofibrosis will be assessed by a blinded assessor who will measure passive and active knee extension and active-assisted knee flexion with a goniometer. For passive knee extension, the patient will lie supine on the examination table with a bolster under the heels with the quadriceps and hamstrings relaxed to assure full passive extension of the knee. For active-assisted knee flexion, the patient will be seated on the examination table with both legs extended and instructed to perform active-assisted knee flexion by placing one hand under their thigh to initiate flexion and then clasp both hands just below the tibial tuberosity. The side-to-side difference in ROM will be determined and interpreted based on IKDC guidelines.
Cost Effectiveness | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months
  Participants who suffer an adverse event will be asked to complete a healthcare resource use diary to capture additional direct and indirect healthcare resources from the time of surgery to the end of the study period. This will include any emergency room visits, hospitalizations, family doctor visits, additional outpatient clinic visits, tests, procedures, prescription or over-the-counter medications and any miscellaneous costs related to their knee. Employment status and time-off paid employment, homemaking or volunteer activities, for both participants and their caregivers, if applicable will be recorded. Quality-adjusted life years (QALYs) using the European Quality of Life Scale (Euro-QoL) will be measured.

IPD SHARING:
Plan to Share IPD: No